CLINICAL TRIAL: NCT00005160
Title: Epidemiology of Cardiovascular Risk Factors in Women (Healthy Women Study)
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1032; R01HL028266-26 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Depression; Carotid Artery Diseases; Menopausal Syndrome
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Depression; Carotid Artery Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and serum samples from baseline and follow up exams stored at -80 degrees Celsius in the Department of Epidemiology, Graduate School of Public Health, University of Pittsburgh.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To determine cardiovascular risk factors and the change in risk factors during and following the menopause.

DETAILED DESCRIPTION:
BACKGROUND:

In 1983, when the Healthy Women Study began, there was a paucity of epidemiological studies of cardiovascular risk factor changes and risk of heart disease related to natural menopause. The Healthy Women Study was one of the few in which the status of premenopausal women was followed carefully through and subsequent to the menopause. The study also included detailed behavioral and biological measures, as well as important environmental factors related to the determinants of these risk factors.

DESIGN NARRATIVE:

A cross-sectional study was conducted to determine the relationship between risk factors, behavioral, psychosocial, and other environmental determinants. A five year longitudinal follow-up of the women evaluated changes over time in risk factors related to the perimenopausal and postmenopausal periods. Longitudinal follow-up after the menopause continues in order to determine the relationships among changes in behavior, hormones, habits, and risk factors.

The women had home interviews, baseline examinations, follow-up of menstrual cycles, and a six-month self-administered questionnaire. Risk factors studied included behavioral factors, glucose and insulin, obesity, exercise, cigarette smoking, nutrition, lipoproteins, blood pressure, and hormones. Surgical menopause and the use of exogenous hormones were also studied. Although not part of the original protocol, measurements of fat distribution, coagulation factors, apoproteins, sodium-lithium counter-transport, and sodium-hydrogen exchange in platelets were added.

The study was renewed in 1995 to continue follow-up to determine characteristics of changes in risk factors, behavioral/psychological attributes and to determine the relationship between risk factors, and their changes and atherosclerotic plaque and wall thickness. Studies are conducted on the interrelationship of lifestyle and behavioral attributed to sex-steroid hormones and insulin and the level of hormones to atherosclerosis. A determination is made of the association of lifestyle to amount and distribution of body fat measured by DEXA and CT of the abdomen.

The study has been renewed several times and ends in November of 2007.

ELIGIBILITY:
Inclusion criteria: Women had to be premenopausal and have an intact uterus and ovaries

Exclusion criteria: hypertension, diabetes, heart disease, major cancer or stroke

Ages: 20 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study began in 1983-84, baseline age was 48, median age was 47. The first EBT examination was added to the study at the approximate time of the 8th postmenopausal visit in 1992-93. 249 women in this grant period.
Sampling Method: Probability Sample
Enrollment: 532 (Actual)
Dates: Start 1983-04; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Predictors of coronary and aortic calcium and carotid intima media thickness and plaque in postmenopausal women at the fourth follow-up of the study | yearly

CONTACTS AND LOCATIONS:
Overall Officials: Lewis Kuller, Principal Investigator — University of Pittsburgh

REFERENCES:
- [Background] Meilahn E, Ferrell R, Kiss J, Temple A, Green F, Humphries S, Kuller L. Genetic determination of coagulation factor VIIc levels among healthy middle-aged women. Thromb Haemost. 1995 Apr;73(4):623-5. PMID 7495069
- [Background] Matthews KA, Kuller LH, Wing RR, Meilahn EN, Plantinga P. Prior to use of estrogen replacement therapy, are users healthier than nonusers? Am J Epidemiol. 1996 May 15;143(10):971-8. doi: 10.1093/oxfordjournals.aje.a008678. PMID 8629615
- [Background] Walker VR, Dombi GW, Gutai JP, Wade DD, Swartz KH, Liu H, Schroeder RR. Semiautomated method for the quantitation of plasma or sera androstenedione, testosterone, and dihydrotestosterone in population studies. Anal Biochem. 1996 Feb 15;234(2):194-203. doi: 10.1006/abio.1996.0072. PMID 8714598
- [Background] Bromberger JT, Matthews KA. A longitudinal study of the effects of pessimism, trait anxiety, and life stress on depressive symptoms in middle-aged women. Psychol Aging. 1996 Jun;11(2):207-13. doi: 10.1037//0882-7974.11.2.207. PMID 8795049
- [Background] Bromberger JT, Matthews KA. A "feminine" model of vulnerability to depressive symptoms: a longitudinal investigation of middle-aged women. J Pers Soc Psychol. 1996 Mar;70(3):591-8. doi: 10.1037//0022-3514.70.3.591. PMID 8851743
- [Background] Bromberger JT, Matthews KA, Kuller LH, Wing RR, Meilahn EN, Plantinga P. Prospective study of the determinants of age at menopause. Am J Epidemiol. 1997 Jan 15;145(2):124-33. doi: 10.1093/oxfordjournals.aje.a009083. PMID 9006309
- [Background] Evans RW, Sankey SS, Hauth BA, Sutton-Tyrrell K, Kamboh MI, Kuller LH. Effect of sample storage on quantitation of lipoprotein(a) by an enzyme-linked immunosorbent assay. Lipids. 1996 Nov;31(11):1197-203. doi: 10.1007/BF02524295. PMID 8934453
- [Background] Lassila HC, Tyrrell KS, Matthews KA, Wolfson SK, Kuller LH. Prevalence and determinants of carotid atherosclerosis in healthy postmenopausal women. Stroke. 1997 Mar;28(3):513-7. doi: 10.1161/01.str.28.3.513. PMID 9056604
- [Background] D'Elio MA, Ness RB, Matthews KA, Kuller LH. Are life stress and social support related to parity in women? Behav Med. 1997 Summer;23(2):87-94. doi: 10.1080/08964289709596732. PMID 9309348
- [Background] Meilahn EN, Kuller LH, Stein EA, Caggiula AW, Matthews KA. Characteristics associated with apoprotein and lipoprotein lipid levels in middle-aged women. Arteriosclerosis. 1988 Sep-Oct;8(5):515-20. doi: 10.1161/01.atv.8.5.515. PMID 3142451
- [Background] Egeland GM, Matthews KA, Kuller LH, Kelsey SF. Characteristics of noncontraceptive hormone users. Prev Med. 1988 Jul;17(4):403-11. doi: 10.1016/0091-7435(88)90039-4. PMID 3217373
- [Background] Matthews KA, Kelsey SF, Meilahn EN, Kuller LH, Wing RR. Educational attainment and behavioral and biologic risk factors for coronary heart disease in middle-aged women. Am J Epidemiol. 1989 Jun;129(6):1132-44. doi: 10.1093/oxfordjournals.aje.a115235. PMID 2729252
- [Background] Wing RR, Bunker CH, Kuller LH, Matthews KA. Insulin, body mass index, and cardiovascular risk factors in premenopausal women. Arteriosclerosis. 1989 Jul-Aug;9(4):479-84. doi: 10.1161/01.atv.9.4.479. PMID 2665702
- [Background] Matthews KA, Meilahn E, Kuller LH, Kelsey SF, Caggiula AW, Wing RR. Menopause and risk factors for coronary heart disease. N Engl J Med. 1989 Sep 7;321(10):641-6. doi: 10.1056/NEJM198909073211004. PMID 2488072
- [Background] Wing RR, Kuller LH, Bunker C, Matthews K, Caggiula A, Meihlan E, Kelsey S. Obesity, obesity-related behaviors and coronary heart disease risk factors in black and white premenopausal women. Int J Obes. 1989;13(4):511-9. PMID 2793303
- [Background] Owens JF, Matthews KA, Wing RR, Kuller LH. Physical activity and cardiovascular risk: a cross-sectional study of middle-aged premenopausal women. Prev Med. 1990 Mar;19(2):147-57. doi: 10.1016/0091-7435(90)90016-d. PMID 2359739
- [Background] Matthews KA, Wing RR, Kuller LH, Meilahn EN, Kelsey SF, Costello EJ, Caggiula AW. Influences of natural menopause on psychological characteristics and symptoms of middle-aged healthy women. J Consult Clin Psychol. 1990 Jun;58(3):345-51. doi: 10.1037//0022-006x.58.3.345. PMID 2365898
- [Background] Kuller LH, Gutai JP, Meilahn E, Matthews KA, Plantinga P. Relationship of endogenous sex steroid hormones to lipids and apoproteins in postmenopausal women. Arteriosclerosis. 1990 Nov-Dec;10(6):1058-66. doi: 10.1161/01.atv.10.6.1058. PMID 2123088
- [Background] Egeland GM, Kuller LH, Matthews KA, Kelsey SF, Cauley J, Guzick D. Hormone replacement therapy and lipoprotein changes during early menopause. Obstet Gynecol. 1990 Nov;76(5 Pt 1):776-82. doi: 10.1097/00006250-199011000-00010. PMID 2170887
- [Background] Wing RR, Matthews KA, Kuller LH, Meilahn EN, Plantinga PL. Weight gain at the time of menopause. Arch Intern Med. 1991 Jan;151(1):97-102. PMID 1985614
- [Background] Meilahn EN, Kuller LH, Matthews KA, Kiss JE. Hemostatic factors according to menopausal status and use of hormone replacement therapy. Ann Epidemiol. 1992 Jul;2(4):445-55. doi: 10.1016/1047-2797(92)90094-7. PMID 1342295
- [Background] Wing RR, Matthews KA, Kuller LH, Smith D, Becker D, Plantinga PL, Meilahn EN. Environmental and familial contributions to insulin levels and change in insulin levels in middle-aged women. JAMA. 1992 Oct 14;268(14):1890-5. PMID 1404713
- [Background] Wing RR. Obesity and weight gain during adulthood: a health problem for United States women. Womens Health Issues. 1992 Summer;2(2):114-20; discussion 120-2. doi: 10.1016/s1049-3867(05)80279-8. No abstract available. PMID 1617307
- [Background] Owens JF, Matthews KA, Wing RR, Kuller LH. Can physical activity mitigate the effects of aging in middle-aged women? Circulation. 1992 Apr;85(4):1265-70. doi: 10.1161/01.cir.85.4.1265. PMID 1555270
- [Background] Matthews KA. Myths and realities of the menopause. Psychosom Med. 1992 Jan-Feb;54(1):1-9. doi: 10.1097/00006842-199201000-00001. PMID 1553395
- [Background] Markovitz JH, Matthews KA, Wing RR, Kuller LH, Meilahn EN. Psychological, biological and health behavior predictors of blood pressure changes in middle-aged women. J Hypertens. 1991 May;9(5):399-406. doi: 10.1097/00004872-199105000-00003. PMID 1649859
- [Background] Costello EJ. Married with children: predictors of mental and physical health in middle-aged women. Psychiatry. 1991 Aug;54(3):292-305. doi: 10.1080/00332747.1991.11024558. PMID 1946829
- [Background] Burgio KL, Matthews KA, Engel BT. Prevalence, incidence and correlates of urinary incontinence in healthy, middle-aged women. J Urol. 1991 Nov;146(5):1255-9. doi: 10.1016/s0022-5347(17)38063-1. PMID 1942274
- [Background] Wing RR, Matthews KA, Kuller LH, Meilahn EN, Plantinga P. Waist to hip ratio in middle-aged women. Associations with behavioral and psychosocial factors and with changes in cardiovascular risk factors. Arterioscler Thromb. 1991 Sep-Oct;11(5):1250-7. doi: 10.1161/01.atv.11.5.1250. PMID 1911710
- [Background] Meilahn EN, Kuller LH, Matthews KA, Wing RR, Caggiula AW, Stein EA. Potential for increasing high-density lipoprotein cholesterol, subfractions HDL2-C and HDL3-C, and apoprotein AI among middle-age women. Prev Med. 1991 Jul;20(4):462-73. doi: 10.1016/0091-7435(91)90044-5. PMID 1908079
- [Background] Egeland GM, Kuller LH, Matthews KA, Kelsey SF, Cauley J, Guzick D. Premenopausal determinants of menopausal estrogen use. Prev Med. 1991 May;20(3):343-9. doi: 10.1016/0091-7435(91)90033-z. PMID 1862056
- [Background] Bunker CH, Wing RR, Mallinger AG, Becker DJ, Matthews KA, Kuller LH. Cross-sectional and longitudinal relationship of sodium-lithium countertransport to insulin, obesity and blood pressure in healthy perimenopausal women. J Hum Hypertens. 1991 Oct;5(5):381-92. PMID 1770468
- [Background] Ickovics JR, Morrill AC, Meisler AW, Rodin J, Bromberger JT, Matthews KA. Employment and coronary risk in women at midlife: a longitudinal analysis. Am J Epidemiol. 1996 Jan 15;143(2):144-50. doi: 10.1093/oxfordjournals.aje.a008723. PMID 8546115
- [Background] Everson SA, Matthews KA, Guzick DS, Wing RR, Kuller LH. Effects of surgical menopause on psychological characteristics and lipid levels: the Healthy Women Study. Health Psychol. 1995 Sep;14(5):435-43. doi: 10.1037//0278-6133.14.5.435. PMID 7498115
- [Background] Davis MC, Matthews KA, Meilahn EN, Kiss JE. Are job characteristics related to fibrinogen levels in middle-aged women? Health Psychol. 1995 Jul;14(4):310-8. doi: 10.1037//0278-6133.14.4.310. PMID 7556034
- [Background] Matthews KA, Kuller LH, Wing RR, Meilahn EN. Biobehavioral aspects of menopause: lessons from the Healthy Women Study. Exp Gerontol. 1994 May-Aug;29(3-4):337-42. doi: 10.1016/0531-5565(94)90013-2. PMID 7925753
- [Background] Cauley JA, Eichner JE, Kamboh MI, Ferrell RE, Kuller LH. Apo E allele frequencies in younger (age 42-50) vs older (age 65-90) women. Genet Epidemiol. 1993;10(1):27-34. doi: 10.1002/gepi.1370100104. PMID 8472931
- [Background] Massoudi MS, Meilahn EN, Orchard TJ, Foley TP Jr, Kuller LH, Costantino JP, Buhari AM. Prevalence of thyroid antibodies among healthy middle-aged women. Findings from the thyroid study in healthy women. Ann Epidemiol. 1995 May;5(3):229-33. doi: 10.1016/1047-2797(94)00110-f. PMID 7606312
- [Background] Kuller LH, Matthews KA, Sutton-Tyrrell K, Edmundowicz D, Bunker CH. Coronary and aortic calcification among women 8 years after menopause and their premenopausal risk factors : the healthy women study. Arterioscler Thromb Vasc Biol. 1999 Sep;19(9):2189-98. doi: 10.1161/01.atv.19.9.2189. PMID 10479662
- [Background] Raikkonen K, Matthews KA, Kuller LH. Anthropometric and psychosocial determinants of visceral obesity in healthy postmenopausal women. Int J Obes Relat Metab Disord. 1999 Aug;23(8):775-82. doi: 10.1038/sj.ijo.0800917. PMID 10490776
- [Background] Raikkonen K, Matthews KA, Kuller LH, Reiber C, Bunker CH. Anger, hostility, and visceral adipose tissue in healthy postmenopausal women. Metabolism. 1999 Sep;48(9):1146-51. doi: 10.1016/s0026-0495(99)90129-4. PMID 10484055
- [Background] Owens JF, Matthews KA. Sleep disturbance in healthy middle-aged women. Maturitas. 1998 Sep 20;30(1):41-50. doi: 10.1016/s0378-5122(98)00039-5. PMID 9819782
- [Background] Matthews KA, Owens JF, Kuller LH, Sutton-Tyrrell K, Lassila HC, Wolfson SK. Stress-induced pulse pressure change predicts women's carotid atherosclerosis. Stroke. 1998 Aug;29(8):1525-30. doi: 10.1161/01.str.29.8.1525. PMID 9707187
- [Background] Simkin-Silverman LR, Wing RR, Plantinga P, Matthews KA, Kuller LH. Lifetime weight cycling and psychological health in normal-weight and overweight women. Int J Eat Disord. 1998 Sep;24(2):175-83. doi: 10.1002/(sici)1098-108x(199809)24:23.0.co;2-b. PMID 9697016
- [Background] Sutton-Tyrrell K, Lassila HC, Meilahn E, Bunker C, Matthews KA, Kuller LH. Carotid atherosclerosis in premenopausal and postmenopausal women and its association with risk factors measured after menopause. Stroke. 1998 Jun;29(6):1116-21. doi: 10.1161/01.str.29.6.1116. PMID 9626281
- [Background] Sutton-Tyrrell K, Kuller LH, Edmundowicz D, Feldman A, Holubkov R, Givens L, Matthews KA. Usefulness of electron beam tomography to detect progression of coronary and aortic calcium in middle-aged women. Am J Cardiol. 2001 Mar 1;87(5):560-4. doi: 10.1016/s0002-9149(00)01431-4. PMID 11230839
- [Background] Kuller LH, Sutton-Tyrrell K, Matthews KA. Blood pressure levels and measurement of subclinical vascular disease. J Hypertens Suppl. 1999 Dec;17(5):S15-9. PMID 10706320
- [Background] Gallo LC, Matthews KA, Kuller LH, Sutton-Tyrrell K, Edmundowicz D. Educational attainment and coronary and aortic calcification in postmenopausal women. Psychosom Med. 2001 Nov-Dec;63(6):925-35. doi: 10.1097/00006842-200111000-00011. PMID 11719631
- [Background] Barinas-Mitchell E, Cushman M, Meilahn EN, Tracy RP, Kuller LH. Serum levels of C-reactive protein are associated with obesity, weight gain, and hormone replacement therapy in healthy postmenopausal women. Am J Epidemiol. 2001 Jun 1;153(11):1094-101. doi: 10.1093/aje/153.11.1094. PMID 11390329
- [Background] Sutton-Tyrrell K, Kuller LH, Matthews KA, Holubkov R, Patel A, Edmundowicz D, Newman A. Subclinical atherosclerosis in multiple vascular beds: an index of atherosclerotic burden evaluated in postmenopausal women. Atherosclerosis. 2002 Feb;160(2):407-16. doi: 10.1016/s0021-9150(01)00591-3. PMID 11849665
- [Background] Mackey RH, Kuller LH, Sutton-Tyrrell K, Evans RW, Holubkov R, Matthews KA. Lipoprotein subclasses and coronary artery calcium in postmenopausal women from the healthy women study. Am J Cardiol. 2002 Oct 17;90(8A):71i-76i. doi: 10.1016/s0002-9149(02)02636-x. PMID 12419483
- [Background] Raikkonen K, Matthews KA, Kuller LH. The relationship between psychological risk attributes and the metabolic syndrome in healthy women: antecedent or consequence? Metabolism. 2002 Dec;51(12):1573-7. doi: 10.1053/meta.2002.36301. PMID 12489070
- [Background] Owens JF, Matthews KA, Raikkonen K, Kuller LH. It is never too late: change in physical activity fosters change in cardiovascular risk factors in middle-aged women. Prev Cardiol. 2003 Winter;6(1):22-8. doi: 10.1111/j.1520-037x.2003.00972.x. PMID 12624558
- [Background] Gallo LC, Troxel WM, Matthews KA, Jansen-McWilliams L, Kuller LH, Sutton-Tyrrell K. Occupation and subclinical carotid artery disease in women: are clerical workers at greater risk? Health Psychol. 2003 Jan;22(1):19-29. PMID 12558198
- [Background] Gallo LC, Troxel WM, Kuller LH, Sutton-Tyrrell K, Edmundowicz D, Matthews KA. Marital status, marital quality, and atherosclerotic burden in postmenopausal women. Psychosom Med. 2003 Nov-Dec;65(6):952-62. doi: 10.1097/01.psy.0000097350.95305.fe. PMID 14645772
- [Background] Gallo LC, Troxel WM, Matthews KA, Kuller LH. Marital status and quality in middle-aged women: Associations with levels and trajectories of cardiovascular risk factors. Health Psychol. 2003 Sep;22(5):453-63. doi: 10.1037/0278-6133.22.5.453. PMID 14570528
- [Background] Harris KF, Matthews KA, Sutton-Tyrrell K, Kuller LH. Associations between psychological traits and endothelial function in postmenopausal women. Psychosom Med. 2003 May-Jun;65(3):402-9. doi: 10.1097/01.psy.0000035720.08842.9f. PMID 12764213
- [Background] Matthews KA, Raikkonen K, Sutton-Tyrrell K, Kuller LH. Optimistic attitudes protect against progression of carotid atherosclerosis in healthy middle-aged women. Psychosom Med. 2004 Sep-Oct;66(5):640-4. doi: 10.1097/01.psy.0000139999.99756.a5. PMID 15385685
- [Background] Mackey RH, Kuller LH, Sutton-Tyrrell K, Evans RW, Holubkov R, Matthews KA. Hormone therapy, lipoprotein subclasses, and coronary calcification: the Healthy Women Study. Arch Intern Med. 2005 Mar 14;165(5):510-5. doi: 10.1001/archinte.165.5.510. PMID 15767525
- [Background] Patel AS, Mackey RH, Wildman RP, Thompson T, Matthews K, Kuller L, Sutton-Tyrrell K. Cardiovascular risk factors associated with enlarged diameter of the abdominal aortic and iliac arteries in healthy women. Atherosclerosis. 2005 Feb;178(2):311-7. doi: 10.1016/j.atherosclerosis.2004.08.026. PMID 15694939
- [Background] Troxel WM, Matthews KA, Gallo LC, Kuller LH. Marital quality and occurrence of the metabolic syndrome in women. Arch Intern Med. 2005 May 9;165(9):1022-7. doi: 10.1001/archinte.165.9.1022. PMID 15883241
- [Background] Park HA, Lee JS, Kuller LH. Relationship between premenopausal dietary intake and postmenopausal subclinical atherosclerosis. Atherosclerosis. 2006 Jun;186(2):420-7. doi: 10.1016/j.atherosclerosis.2005.08.002. Epub 2005 Sep 22. PMID 16182299
- [Background] Gianaros PJ, Salomon K, Zhou F, Owens JF, Edmundowicz D, Kuller LH, Matthews KA. A greater reduction in high-frequency heart rate variability to a psychological stressor is associated with subclinical coronary and aortic calcification in postmenopausal women. Psychosom Med. 2005 Jul-Aug;67(4):553-60. doi: 10.1097/01.psy.0000170335.92770.7a. PMID 16046367